CLINICAL TRIAL: NCT06827444
Title: Effects of Attention and Placebo Modulation on Cycling Performance: an Experimental Study on Stationary Bikes
Brief Title: The Role of Attention in Modulating the Placebo Effect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesco Pagnini, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Università Cattolica del Sacro
Record Dates: First submitted 2024-06-27; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Placebo Effect; Attention
Keywords: Placebo; Bayesiana approach; Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo
- Control Group (Active Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Participants will be provided with a chest strap for heart rate measurement (the strap will be washed and disinfected after each session), connected to the Polar Beat app downloaded by the researcher. Subsequently, each participant will perform an initial 10-minute baseline warm-up session (a cadence of 70-80 RPM will be requested). From the cycle ergometer display, values for watts (the amount of work done per second), power (the amount of work done over a certain period of time), and speed (expressed in kilometers per hour) will also be extracted. During the test, no visual or verbal feedback will be provided. Participants will be blind to the cycle ergometer screen, so the data will not influence their behavior. Heart rate will be continuously recorded throughout the exercise period and during the participant's recovery. Participants will then be randomized to one of the following manipulations.

SUMMARY:
This project aims to examine whether these forms of attention to sensory information can modulate the mind-body interaction. This will be demonstrated through a study focused on the placebo effect with attention manipulation. Specifically, the project will focus on the construct of mindful attention to increase the precision of the likelihood and reduce the effects of priors, and on directed attention to modify the position and precision of the likelihood, hypothetically modulating the placebo effect.

The study involves recruiting 128 healthy individuals, who will be asked to cycle on an ergometer for approximately 60 minutes, with alternating phases in which attention will be manipulated. After an initial warm-up phase, they will receive a placebo drink, presented as "highly stimulating." An additional group of 32 participants will not receive either the placebo drink or the attentional stimuli, but will undergo the same training cycles. All participants will receive a pre-intervention assessment, and heart rate, emotions, and perceived fatigue will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Persons (18+) in good health, verified by presenting a medical certificate (sporting, competitive or non-competitive, or of good health).
* Be available to go to a gym. If not enrolled, the cost of admission is borne by the project.

Exclusion Criteria:

* known cardiovascular diseases, gastrointestinal diseases, musculoskeletal injuries, upper respiratory tract infections;
* allergy and/or intolerance to caffeine.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 30 minutes
  Numeric Rating Scale 0-10, where 10 indicates maximum fatigue.

SECONDARY OUTCOMES:
Heart rate | 30 minutes
  Heart rate beats, assessed with Polar H10 chest strap
Perceived efficacy of the energy drink | 30 minutes
  Numeric Rating Scale 0-10, where 10 is the most effective.

OTHER OUTCOMES:
Mindfulness | Once, at the baseline (pre-experiment)
  The Mindfulness Awareness Attention Scale (MAAS) is a widely used self-report measure designed to assess an individual's level of mindfulness, particularly focusing on present-moment awareness and attention. Developed by MacKillop and Anderson (2007), the scale evaluates the frequency of mindful states in everyday life, emphasizing the ability to remain attentive to and aware of current experiences. The MAAS has been extensively applied in both clinical and non-clinical settings to explore the relationship between mindfulness and various psychological and behavioral outcomes, such as stress reduction, emotional regulation, and overall well-being.
Anxiety | Once, at the baseline (pre-experiment)
  The Beck Anxiety Inventory (BAI) is a widely used self-report measure designed to assess the severity of anxiety symptoms. Developed by Beck et al. (1988), the scale focuses on somatic and subjective symptoms of anxiety, such as nervousness, fear, and physical sensations like sweating or dizziness. The BAI is commonly used in both clinical and research settings to screen for anxiety disorders, monitor symptom changes over time, and evaluate the effectiveness of therapeutic interventions. Its reliability and ease of use make it a valuable tool for assessing anxiety across diverse populations.
Stress | Once, at the baseline (pre-experiment)
  The Perceived Stress Scale (PSS) is a widely used self-report tool designed to measure the level of stress an individual perceives in their daily life. Developed by Cohen et al. (1994), the scale evaluates how unpredictable, uncontrollable, and overwhelming respondents find their life circumstances over the past month. The PSS is often employed in both research and clinical settings to assess stress levels, explore its impact on health outcomes, and monitor changes following interventions aimed at stress reduction. Its versatility and simplicity make it suitable for diverse populations and contexts.
Optimism | Once, at the baseline (pre-experiment)
  The Life Orientation Test - Revised (LOT-R) is a psychological assessment tool designed to measure individual differences in dispositional optimism. Developed by Scheier et al. (1994), the LOT-R evaluates the extent to which individuals hold positive expectations about future outcomes. This self-report scale is widely used in both research and clinical settings to examine the role of optimism in psychological well-being, health outcomes, and coping strategies. Its concise format and strong psychometric properties make it a valuable instrument for exploring optimism across various populations and contexts.
Cognitive flexibility | Once, at the baseline (pre-experiment)
  The Cognitive Flexibility Scale (CFS) is a self-report instrument designed to assess an individual's capacity to adapt their thinking and behavior in response to changing situations or environments. Developed by Martin and Rubin (1995), the scale evaluates key aspects of cognitive flexibility, including the ability to consider multiple perspectives, generate alternative solutions, and cope effectively with challenges. This tool is widely used in research and clinical settings to explore how cognitive flexibility influences problem-solving, resilience, and overall psychological well-being. Its straightforward design ensures usability across diverse populations.
Personality traits | Once, at the baseline (pre-experiment)
  The Big Five Inventory-10 (BFI-10) is a brief self-report measure designed to assess the five major dimensions of personality: openness, conscientiousness, extraversion, agreeableness, and neuroticism. Developed as a shortened version of the original Big Five Inventory, it includes only 10 items, making it ideal for contexts where time is limited, while still providing reliable and valid results (Rammstedt & John, 2007). Despite its brevity, the BFI-10 retains the ability to capture key personality traits and is widely used in psychological research and applied settings to gain insights into individual differences.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca NA Grosso, MD, Study Director — Catholic University of the Sacred Heart
Locations (1):
- Università Cattolica del Sacro Cuore, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No